CLINICAL TRIAL: NCT00723320
Title: Effect of Atorvastatin and Lifestyle Intervention on Progression of Carotid Intima-Media Thickness in Chinese People Without Manifest Atherosclerotic Disease
Brief Title: Effect of Atorvastatin and Lifestyle Intervention on Progression of Pre-Clinical Atherosclerosis
Acronym: EALIPPCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Collaborators: Peking University First Hospital (Other)
Responsible Party: Yong Huo, Peking University First Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 2006BAI01A02-03
Record Dates: First submitted 2008-07-21; First posted 2008-07-28 (Estimated); Last update posted 2008-08-25 (Estimated); Status verified 2008-07

CONDITIONS: Atherosclerosis
Keywords: Atherosclerosis; Atorvastatin; Therapeutic lifestyle change; CIMT; ABI; PWV
MeSH Terms: conditions — Atherosclerosis | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- P+N (No Intervention): placebo without lifestyle intervention
- D+N (Experimental): Atorvastatin 10mg/d
  Interventions: Drug: Atorvastatin
- P+A (Experimental): lifestyle intervention without Atorvastatin
  Interventions: Behavioral: Aggressive lifestyle intervention
- D+A (Experimental): lifestyle intervention and Atorvastatin 10mg/d
  Interventions: Drug: Atorvastatin; Behavioral: Aggressive lifestyle intervention

INTERVENTIONS:
Drug: Atorvastatin — atorvastatin 10mg/d
  Arms: D+A; D+N
Behavioral: Aggressive lifestyle intervention — aggressive lifestyle intervention
  Arms: D+A; P+A

SUMMARY:
The purpose of this study is to determine whether atorvastatin, aggressive lifestyle intervention, and their interaction are effective in delaying the progress of pre-clinical atherosclerosis.

DETAILED DESCRIPTION:
Primary prevention of atherosclerotic disease remains a big challenge. Currently, it is not clear how to treat those subjects with evidence of pre-clinical atherosclerosis but without obvious conventional risk factors. This randomized, placebo controlled, double blind study is to evaluate the effect of Atorvastatin 10 mg daily, therapeutic lifestyle change, and their combination, on the progression of CIMT in those with higher baseline CIMT value but are not belong to 'high risk' category, according to the conventional risk factors.

ELIGIBILITY:
Inclusion Criteria:

* CIMT is not less than 0.9 mm
* without Clinical diagnosis of atherosclerotic disease
* without Diabetes

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2008-02; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
The progress of CIMT | 2 years

SECONDARY OUTCOMES:
The progress of ABI | 2 years
The progress of PWV | 2 years
Occurrence of atherosclerotic disease | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Li, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China